CLINICAL TRIAL: NCT04033770
Title: Assessment of the Lower Urinary Tract: Consistency, Features and Artifacts of Invasive Urodynamic Assessments - a Randomized Controlled Trial
Brief Title: Urodynamic Assessment of the Lower Urinary Tract: Water vs. Air
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: UDI-RCT 2018-00073
Record Dates: First submitted 2019-03-26; First posted 2019-07-26 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2022-02

CONDITIONS: Lower Urinary Tract Dysfunction
Keywords: Urodynamic investigation; Lower urinary tract dysfunction; Water-perfused catheter; Air-charged catheter

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Air-charged measurement system (Active Comparator): UDI (same session repeat filling cystometry and pressure flow study) according to "Good Urodynamic Practice" recommended by the ICS but using an air-charged instead of a water-filled measurement system.
  Interventions: Other: Urodynamic investigation
- Water-perfused measurement system (Active Comparator): UDI (same session repeat filling cystometry and pressure flow study) according to "Good Urodynamic Practice" recommended by the ICS.
  Interventions: Other: Urodynamic investigation

INTERVENTIONS:
Other: Urodynamic investigation — Urodynamic investigation using an air-charged measurement system
  Arms: Air-charged measurement system
Other: Urodynamic investigation — Urodynamic investigation using a water-perfused measurement system
  Arms: Water-perfused measurement system

SUMMARY:
Comparison of water-perfused (WP) and air-charged (AC) catheters for invasive urodynamic investigation (UDI) regarding consistency, features and artifacts.

DETAILED DESCRIPTION:
UDI is the gold standard to assess refractory lower urinary tract symptoms (LUTS), i.e. to detect and specify lower urinary tract dysfunction (LUTD). Therefore, UDI findings lead to diagnosis and decision-making for further non-invasive and invasive therapies. For UDI pressure recordings, the use of WP catheters is recommended by the International Continence Society (ICS).

Currently AC catheters have been marked for pressure recording as an alternative to WP catheters. However, the number of comparative studies is very limited. Nevertheless, since release, AC catheters have gained popularity due to their omnidirectional detection of pressure, and claimed reduction in movement artefacts (due to weight-less air column vs weighted water column), lack of external reference level, and ease of set-up/use. Still, there is debate whether AC catheters are an acceptable alternative to fluid-filled lines for measuring intravesical and intra-abdominal pressure in UDI. Based on the available literature, an appropriate conclusion, whether both systems can be used as equivalents and interchangeably, cannot be drawn.

In this study we compare both systems regarding consistency, features and artifacts.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients with LUTD
* Age: minimum 18 years
* Informed consent
* Competent German language skills

Exclusion Criteria:

* Age <18 years
* Pregnancy or breast feeding (see chapter 3.6.)
* Symptomatic UTI
* Individuals especially in need of protection
* No informed consent
* Patients incapable to follow the trial, e.g. because of language problems, psychiatric disorders, dementia and so on.
* Earlier participation in this clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 490 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-02-11 (Actual); Study Completion 2022-02-11 (Actual)

PRIMARY OUTCOMES:
Artefact susceptibility of the measurement systems | During the urodynamic investigation
  Number of Artifacts impairing the quality/interpretability of the urodynamic examination

SECONDARY OUTCOMES:
Subjective perception of pain and discomfort (on a visual analog scale) between the measurement systems | During the urodynamic investigation
  Perception of pain and discomfort on a visual analog scale (presented as a 100-mm horizontal line on which the patient's pain and discomfort intensity is represented by a point between the extremes of "no pain/discomfort at all" and "worst pain/discomfort imaginable (from 0 to 10))
Incidence of side effects: number and intensity/severity (mild/moderate/severe) of AEs and SAE for the following categories during and for 7 days after the urodynamic investigation using an air-charged vs. water-perfused measurement system | Once during urodynamic investigation and 7 days thereafter
  Infection - Urinary Tract Infection (UTI); severe or sudden increase in pain; severe or sudden increase in spasticity; autonomic dysreflexia; urgent (unexpected) transfer/admittance to an acute care facility
Difference in volumetric during urodynamic investigation using an air-charged vs. water-perfused measurement system | During the urodynamic investigation
  Cystometric capacity [mL], volume at first DO [mL], voided volume [mL] and post void residual [mL] as assessed by urodynamic measurement
Difference in Compliance [mL/cmH2O] during urodynamic investigation using an air-charged vs. water-perfused measurement system | During the urodynamic investigation
Difference in Pressure changes during urodynamic investigation using an air-charged vs. water-perfused measurement system | During the urodynamic investigation
  Maximum DO amplitude [cmH2O], detrusor leak-point pressure [cmH2O], maximum detrusor pressure [cmH2O] during storage phase, maximum detrusor pressure [cmH2O] during voiding phase, detrusor pressure at maximum flow rate [cmH2O]
Difference in in maximum flow rate [mL/s] during urodynamic investigation using an air-charged vs. water-perfused measurement system | During the urodynamic investigation

CONTACTS AND LOCATIONS:
Locations (1):
- Universitätsklinik Balgrist, Zurich, Switzerland